CLINICAL TRIAL: NCT00245375
Title: A Randomized Controlled Trial Comparing Combination Therapy of Acetaminophen Plus Ibuprofen Versus Tylenol #3 for the Treatment of Pain After Outpatient Surgery
Brief Title: A Trial Comparing Combination Therapy of Acetaminophen Plus Ibuprofen Versus Tylenol #3 for the Treatment of Pain After Outpatient Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDHA003
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Laparoscopic Cholecystectomy; Inguinal Hernia; Abdominal Hernia; Umbilical Hernia
Keywords: Outpatient Surgery for:; inguinal hernia repair; abdominal hernia repair; umbilical hernia repair
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Abdominal; Hernia, Umbilical | interventions — Acetaminophen; Ibuprofen

INTERVENTIONS:
Drug: Tylenol #3
Drug: Combination Tylenol and Ibuprofen

SUMMARY:
Increasingly in general surgery, the investigators are conducting outpatient day surgery. Ambulatory surgery currently comprises 60 to 70% of surgeries performed in North America. These patients all require some form of analgesia which can be taken at home in the first few days after the surgery. The current standard at the investigators' centre and many others in the maritime provinces is to provide a prescription for oral acetaminophen plus codeine or oxycodone (Tylenol #3®, Percocet ®). Some patients may receive more potent opioids such as oral hydromorphone (Dilaudid®). Unfortunately, the most commonly prescribed medication (Tylenol #3®) is often poorly tolerated by patients, has several undesirable side effects, and may not provide effective pain relief. In the investigators' experience, non-steroidal anti-inflammatory drugs (NSAIDs) are uncommonly a routine addition to the home analgesic regimen.

Tylenol #3®, in the investigators' experience and opinion, is a poor post surgical pain medication. They hope to show that a combination of ibuprofen and acetaminophen is better for pain relief after these procedures. The combination of acetaminophen and ibuprofen would be a safe, cheap, and readily available regimen. Unfortunately, as the prescribing practices of surgeons are old habits, it will require a very convincing argument to get them to change their practices. A randomized controlled trial comparing these two regimens, the investigators hope, would be a powerful enough argument.

The hypothesis of this study, therefore, is that the pain control provided by a combination of acetaminophen plus ibuprofen (650 mg/400 mg four times per day) will be superior to Tylenol #3® (600 mg acetaminophen/60 mg codeine/15 mg caffeine four times per day).

This study will attempt to enroll 150 patients in total. Eligible patients will be identified by their attending surgeon and contacted by study personnel. Patients who enroll in the study will undergo their surgery in the usual manner. After the surgery, in the recovery room, once they are ready to go home, they will be randomized to receive combination A or B and be given a week's worth of pain medication. They will then go home and take this medication as directed. They will record their pain intensity and pain relief once per day using a diary provided in the study package. One week after their surgery, they will return to the hospital clinic and be seen by the study nurse. They will hand over the diary and any unused medication. They will also be asked several questions regarding their overall satisfaction, incidence of side effects, and how long until they were pain free.

The risks of participating in this study are minimal from the risks inherent to the procedures and medications the patients would receive within the standard of care. Ibuprofen is a commonly used NSAID which is widely available over the counter and has an established safety profile. The most common adverse effects of ibuprofen and other NSAIDs are gastrointestinal bleeding and ulceration. Other less common adverse effects include nephrotoxicity, hypersensitivity reactions, hepatic dysfunction (longterm use), and cognitive dysfunction. The investigators' patients will be selected to exclude those most at risk for these complications (see exclusion criteria). Acetaminophen has few side effects, with no adverse effects on platelet function and no evidence of gastric irritation.

ELIGIBILITY:
Inclusion Criteria:

Patients may take part in this study if the answer is YES to all of these questions:

* Female or male between 17-65 years of age
* Going to have one of the following surgeries:

  * umbilical hernia repair
  * inguinal hernia repair
  * small incisional or abdominal wall hernia repair
  * laparoscopic cholecystectomy (gallbladder removed)
* Going home after their surgery the same day
* Have signed consent form.

Exclusion Criteria:

Patients have had or have:

* Been diagnosed with peptic ulcer disease or bleeding stomach ulcer in the recent past and are not currently on a proton pump inhibitor (special antacid medication, eg. Losec®, Pantoloc®, Prevacid®, Nexium®).
* Suffered from asthma
* Allergies to codeine, non-steroidal anti-inflammatory drugs (Advil®, Ibuprofen), aspirin, or acetaminophen
* Been taking other prescription pain medications prior to their surgery
* A history of chronic pain disorder
* Fibromyalgia (a chronic pain illness with symptoms of muscle aches, pain, stiffness, general fatigue and sleep problems)
* Active kidney disease or failure
* Known liver disease
* Are females who are pregnant or nursing
* A problem with alcohol or drug abuse.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2005-01; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Mean daily and final visual analog scale (VAS) scores
Mean daily and final Likert scores
Total pain relief
Sum of pain intensity differences
Cumulative weekly VAS scores

SECONDARY OUTCOMES:
Treatment failures
Amount of medication used
Days to stopping medication
Incidence of side effects
Compliance with regimen

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey A Porter, MD, FRCSC, Study Director — CDHA/Dalhousie University
Locations (1):
- Dartmouth General Hospital, Dartmouth, Nova Scotia, Canada